CLINICAL TRIAL: NCT03313700
Title: Randomized Controlled Trials on Clinical Outcomes of Robotic Versus Laparoscopic Distal Gastrectomy for Gastric Cancer
Brief Title: Clinical Outcomes of Robotic Versus Laparoscopic Distal Gastrectomy for Gastric Cancer
Acronym: RDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of gastric surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02
Record Dates: First submitted 2017-10-10; First posted 2017-10-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stomach Neoplasm; Robotic Surgery
Keywords: Stomach Neoplasm; Robotic Surgery; Distal Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Distal Gastrectomy (Experimental): Robotic Distal Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Robotic Distal Gastrectomy
- Laparoscopic Distal Gastrectomy (Active Comparator): Laparoscopic Distal Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic Distal Gastrectomy

INTERVENTIONS:
Procedure: Robotic Distal Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case, robotic distal gastrectomy will be performed in the experimental group.
  Arms: Robotic Distal Gastrectomy
Procedure: Laparoscopic Distal Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case, laparoscopic distal gastrectomy will be performed in the comparator group.
  Arms: Laparoscopic Distal Gastrectomy

SUMMARY:
The purpose of this study is to explore the clinical outcomes of the robotic distal gastrectomy for patients with gastric adenocarcinoma（cT1-4a, N-/+, M0）.

DETAILED DESCRIPTION:
Robotic surgery has been developed with the aim of improving surgical quality and overcoming the limitations of conventional laparoscopy in the performance of complex mini-invasive procedures. The study is designed to explore the clinical outcomes of the robotic distal gastrectomy by comparing short- and long-term outcomes including financial cost of robotic and laparoscopic distal gastrectomy in the treatment of gastric adenocarcinoma （cT1-4a, N-/+, M0）.

ELIGIBILITY:
Inclusion Criteria:

1. Age from over 18 to under 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT1-4a(clinical stage tumor), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. expected to perform distal gastrectomy with D1+/D2 lymph node dissction to obtain R0 resection sugicall results.
5. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastric surgery (except ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
5. Gastric multiple primary carcinoma
6. Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
7. History of other malignant disease within the past 5 years
8. History of previous neoadjuvant chemotherapy or radiotherapy
9. History of unstable angina or myocardial infarction within the past 6 months
10. History of cerebrovascular accident within the past 6 months
11. History of continuous systematic administration of corticosteroids within 1 month
12. Requirement of simultaneous surgery for other disease
13. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
14. FEV1<50% of the predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  the rate of 3-year disease free survival

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
  the rate of 3-year overall survival rate
3-year recurrence pattern | 36 months
  the pattern of recurrence in 3 years
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
overall postoperative serious morbidity rates | 30 days
  Refers to the incidence of early postoperative complication which is graded as Clavien-Dindo IIIA or higher
number of retrieved lymph nodes | 1 days
  number of retrieved lymph nodes
the noncompliance rate of lymphadenectomy | 1 days
  the noncompliance rate of lymphadenectomy
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight in kilograms on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
The variation of cholesterol | 3, 6, 9 and 12 months
  The variation of cholesterol in millimole/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
The variation of album | 3, 6, 9 and 12 months
  The variation of album in gram/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
The variation of white blood cell count | Preoperative 7 days and postoperative 1 and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 5 are recorded to access the inflammatory response.
The variation of hemoglobin | Preoperative 7 days and postoperative 1 and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 5 are recorded to access the inflammatory response.
Hospitalization expenses | 30 days
  The cost from admission to discharge
operation time | 1 days
  operation time

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Lu J, Wu D, Huang JB, Lin J, Xu BB, Xue Z, Zheng HL, Lin GS, Shen LL, Li P, Wang JB, Lin JX, Chen QY, Cao LL, Xie JW, Zheng CH, Huang CM. Comparison of robotic versus laparoscopic versus open distal gastrectomy for locally advanced gastric cancer: a prospective trial-based economic evaluation. Surg Endosc. 2023 Oct;37(10):7472-7485. doi: 10.1007/s00464-023-10147-1. Epub 2023 Jul 3. PMID 37395806